CLINICAL TRIAL: NCT00005325
Title: Identifying Genes Involved in Abnormal Blood Pressure - Hypertension SCOR
Status: Completed | Type: Observational
Sponsor: Boston University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4109; P50HL055001 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

SUMMARY:
To seek out genes or genetic markers which identify subjects more vulnerable to hypertension under the influence of environmental factors.

DETAILED DESCRIPTION:
BACKGROUND:

Essential hypertension is a multifactorial disorder with a Gaussian distribution and with a genetic component that appears to be polygenic and heterogeneous. The studies require clinical knowledge of the pathophysiology and therapy of hypertension, availability of a large racially diverse patient population and a General Clinical Research Center for recruitment, characterization and classification of subjects, in combination with knowledge of molecular biology for DNA preparation and expertise in molecular genetics and molecular epidemiology for genetic analysis.

The study is part of a Specialized Centers of Research initiative in the Molecular Genetics of Hypertension. The initiative originated in deliberations of the September 1992 National Heart, Lung, and Blood Advisory Council. In May 1993, a program evaluation committee convened by the NHLBI was charged with the task of assessing the overall goals of the Hypertension SCOR program and of recommending areas of future need. The committee's recommendations formed the basis of this proposed initiative which was released as a Request for Applications in December, 1993.

DESIGN NARRATIVE:

The study, a subproject within a Hypertension Specialized Center of Research (SCOR), had five substudies between 1996 and 2001. The first classified hypertensives into relatively homogeneous subgroups according to intermediate phenotypes based on heritable biological traits, including anthropometric and neurohumoral data obtained by submitting selected subjects to a 3-day inpatient protocol, from which data were extrapolated and applied to stratify larger subject populations in order to enhance efficacy of subsequent genetic analysis. The second substudy genotyped subjects for chromosomal loci using approximately 350 highly polymorphic microsatellite markers spaced every 5-10 centimorgans (cM) along each chromosome. The strategy was to initially type markers in a select group of hypertensive kindreds that independently demonstrated linkage. The third substudy analyzed the genetic marker data for linkage using both parametric (lod score) and nonparametric (affected-pedigree-member) methods. Suggestive findings were pursued in the sib-pairs. The fourth substudy used the case-control method to confirm positive linkage from substudy 3 and to identify particular allele associations using methods of linkage disequilibrium and DNA pooling. The fifth substudy screened and assessed mutations in candidate genes linked to hypertension in patients and controls. A collaboration was established with the Framingham Heart Study, with linkage analyses conducted for hypertension in this cohort.

The subproject was renewed in February 2001 through 2006 to continue the clinical studies and to expand the collection of hypertensive families, including subjects who have undergone extensive clinical evaluation and who can be subgrouped into intermediate phenotypes, as well as families from genetically isolated populations from Greece, Israel, and South Africa. Various subsets of this population will be submitted to different genetic analyses as appropriate, including linkage and association studies, genome-wide scan for genetic isolates, evaluation of single nucleotide polymorphisms in selected genes, testing of quantitative trait loci (QTL) by micro satellite markers and mapping of promising marrow regions by DNA sequencing.

ELIGIBILITY:
No eligibility criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1996-02; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haralambos Gavras — Boston University

REFERENCES:
- [Background] Baima J, Nicolaou M, Schwartz F, DeStefano AL, Manolis A, Gavras I, Laffer C, Elijovich F, Farrer L, Baldwin CT, Gavras H. Evidence for linkage between essential hypertension and a putative locus on human chromosome 17. Hypertension. 1999 Jul;34(1):4-7. doi: 10.1161/01.hyp.34.1.4. PMID 10406815
- [Background] Levy D, DeStefano AL, Larson MG, O'Donnell CJ, Lifton RP, Gavras H, Cupples LA, Myers RH. Evidence for a gene influencing blood pressure on chromosome 17. Genome scan linkage results for longitudinal blood pressure phenotypes in subjects from the framingham heart study. Hypertension. 2000 Oct;36(4):477-83. doi: 10.1161/01.hyp.36.4.477. PMID 11040222
- [Background] Nicolaou M, DeStefano AL, Gavras I, Cupples LA, Manolis AJ, Baldwin CT, Gavras H, Farrer LA. Genetic predisposition to stroke in relatives of hypertensives. Stroke. 2000 Feb;31(2):487-92. doi: 10.1161/01.str.31.2.487. PMID 10657427
- [Background] Erlich PM, Cui J, Chazaro I, Farrer LA, Baldwin CT, Gavras H, DeStefano AL. Genetic variants of WNK4 in whites and African Americans with hypertension. Hypertension. 2003 Jun;41(6):1191-5. doi: 10.1161/01.HYP.0000070025.30572.91. Epub 2003 Apr 28. PMID 12719438
- [Background] Zhou XF, Cui J, DeStefano AL, Chazaro I, Farrer LA, Manolis AJ, Gavras H, Baldwin CT. Polymorphisms in the promoter region of catalase gene and essential hypertension. Dis Markers. 2005;21(1):3-7. doi: 10.1155/2005/487014. PMID 15735318
- [Background] Manolis AJ, Iraklianou S, Pittaras A, Zaris M, Tsioufis K, Psaltiras G, Psomali D, Foussas S, Gavras I, Gavras H. Arterial compliance changes in diabetic normotensive patients after angiotensin-converting enzyme inhibition therapy. Am J Hypertens. 2005 Jan;18(1):18-22. doi: 10.1016/j.amjhyper.2004.08.014. PMID 15691612
- [Background] Cui J, Melista E, Chazaro I, Zhang Y, Zhou X, Manolis AJ, Baldwin CT, Destefano AL, Gavras H. Sequence variation of bradykinin receptors B1 and B2 and association with hypertension. J Hypertens. 2005 Jan;23(1):55-62. doi: 10.1097/00004872-200501000-00013. PMID 15643125